CLINICAL TRIAL: NCT02754713
Title: Prognostic Biomarkers in Patients With Acute Pericarditis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hippocration General Hospital (Other)
Responsible Party: Principal Investigator, George Lazaros, Consultant Cardiologist, Hippocration General Hospital
Other Study IDs: 14167/20/08/2009
Record Dates: First submitted 2016-04-20; First posted 2016-04-28 (Estimated); Last update posted 2016-04-28 (Estimated); Status verified 2016-04

CONDITIONS: Pericarditis
MeSH Terms: conditions — Pericarditis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples will be collected for plasma biomarkers (e.g. circulating pro-inflammatory cytokines, miRNAs etc)
  Image datasets from available imaging tests will be also analysed to quantify imaging biomarkers (e.g. epicardial fat volume from computerised tomography, speckle-tracking analysis for cardiac ultrasound etc.).
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with acute pericarditis: 300 patients with a first episode of acute pericarditis

SUMMARY:
The study will aim at investigating novel plasma or imaging biomarkers in patients with acute pericarditis. All participants will be treated according to established clinical recommendations for the diagnosis and treatment of acute pericarditis.

Study participants will undergo blood sampling for measurements of plasma biomarkers potentially involved in the pathogenesis of acute pericarditis. Imaging datasets from available imaging tests will be used to quantify imaging biomarkers. Patients will be followed up prospectively for up to 18 months. The prognostic value of plasma and/or imaging biomarkers for development of complications such as atrial fibrillation, pericarditis recurrences, constrictive pericarditis and/or the need to switch to 2nd line treatment will be sought.

DETAILED DESCRIPTION:
Background: Acute pericarditis is a relatively common disorder with a reported incidence ranging from 3.32 to 27.7 cases per 100,000 persons per year in the Western word.Potential complications of acute pericarditis include pericarditis recurrence, cardiac tamponade and constrictive pericarditis.To date there is limited clinical evidence on prognostic factors of outcome in acute pericarditis; use of steroids/colchicine, the kinetics of C-reactive protein (CRP) in the acute phase and the underlying aetiology have been previously associated with recurrence of acute pericarditis. Nevertheless there are currently no established biomarkers to risk stratify patients with acute pericarditis.

Methods:

This will be a prospective observational study in three hundred (n=300) patients with a first diagnosis of acute pericarditis to explore the value of plasma or imaging biomarkers in predicting clinical outcome.

Written informed consent will be obtained obtained from all patients. The protocol has been approved by the Institutional Ethics Committee (ref. number 14167/20/08/2009) and will be carried out in accordance with the principles of the declaration of Helsinki.

Diagnosis of acute pericarditis and choice of treatment Acute pericarditis was diagnosed based on clinical recommendations. Baseline clinical and demographic data were recorded in all cases. In line with the current guidelines, diagnostic work-up included clinical history and examination, ECG, chest x-ray, echocardiography and routine blood tests including among others high-sensitivity cardiac troponin I and CRP.12 In patients with high risk features for secondary forms or complicated course13 additional tests will be performed at the discretion of the attending physician.

Ibuprofen 600mg tid or aspirin 1gr tid will be given as first line therapy for at least 7-10 days provided that CRP is normalized within the same time interval, and subsequent tapering in the following 3-4 weeks. Steroids will be given at a dose of 0.2-0.5mg/kg of prednisolone or equivalent dose of another steroid until CRP normalization and symptoms resolution followed by tapering according to recommendations. Indications for steroids administration as a first line treatment included secondary cause of pericarditis and contraindications or poor response to NSAIDs treatment (persisting symptoms and/or CRP elevation beyond 10 days of treatment). Colchicine will be given in all cases at a dose of 0.5mg bid (unless contraindicated) and halved in patients aged >70 years old or body weight <70kg.Treatment failure with first line medication and/or switch to steroids for any reason was recorded.

Clinical follow-up All patients included will be followed-up at outpatients' clinic at 2 weeks, 1 month, 2 months post-hospital discharge and every 3 months thereafter (or earlier if symptomatic) up to a total of 18 months, given that the majority of clinical complications appear within this time frame.The composite clinical end-point will be poor response to NSAIDs treatment (defined by the need to switch to 2nd line therapy) and development of either recurrent, incessant or constrictive pericarditis.

Pericarditis will be diagnosed as incessant if lasting more than 4-6 weeks but less than 3 months and recurrent in the presence of 4-6 weeks symptom-free interval of 4-6 weeks between 2 consecutive episodes.

Measurement of plasma biomarkers The prognostic value of plasma biomarkers such as CRP, troponin I, proinflammatory cytokines (e.g. IL-6, IL18 and others) in patients with acute pericarditis will be investigated. The value of micro-RNAs (miRNAs) as candidate biomarkers involved in the pathogenesis of acute pericarditis will be also sought in gene expression studies.

Measurement of Imaging biomarkers Stored imaging datasets (e.g.cardiac ultrasound images, cardiac computed tomography data etc) will be used to explore the value of imaging biomarkers (e.g epicardial fat volume by computed tomography, speckle-tracking analysis of cardiac ultrasound) in predicting clinical outcome of patients with acute pericarditis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with first diagnosis of acute pericarditis

Exclusion Criteria:

* Not willing to provide written consent

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with first diagnosis of acute pericarditis
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2009-09; Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Development of of constrictive, recurrent or incessant pericarditis or poor response to NSAIDs treatment. | Up to 18 months after hospital discharge
  Participants will be followed-up by scheduled visits at the Outpatients' Clinic at 2 weeks, 1 month, 2 months post-hospital discharge and every 3 months thereafter (or earlier if symptomatic) up to a total of 18 months.

SECONDARY OUTCOMES:
Development of new atrial fibrillation | Development of new atrial fibrillation at 7 days.
  Patients will be monitored by daily ECGs up to 1 week for the development of new atrial fibrillation

CONTACTS AND LOCATIONS:
Overall Officials: Dimitris Tousoulis, Professor, Study Director — Cardiology Department, Hippokration Hospital, Athens Medical School
Locations (1):
- Cardiology Department, Hippokration Hospital, Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: Undecided